CLINICAL TRIAL: NCT00002088
Title: Treatment of Patients With Human Immunodeficiency Virus (HIV)-Related Chronic Diarrhea With Saccharomyces Boulardii or Placebo: A Double Blind Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocodex (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 083A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: Diarrhea; HIV Infections
Keywords: Diarrhea; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Saccharomyces
MeSH Terms: conditions — Diarrhea; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

INTERVENTIONS:
Drug: Saccharomyces boulardii

SUMMARY:
To assess the efficacy of Saccharomyces boulardii (a nonpathogenic yeast) in producing a significant reduction in diarrheal symptoms in HIV-infected patients with chronic diarrhea.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiviral medication for HIV infection.

Patients must have:

* Documented HIV infection.
* Chronic diarrhea (for at least 1 month) that is either a manifestation or complication of documented HIV infection.
* Had a stool culture (Salmonella, Shigella, Campylobacter, and Clostridium difficile) and stool analysis for ova and parasite (O/P X 3) within the past 2 months.
* Failed antimicrobial treatment for diarrhea OR received no prior antimicrobials for stool pathogens because stool cultures were negative.

Patients who are on antiviral medications for HIV infection must have received such medication for at least 2 weeks and must remain on stable dose for weeks 1 and 2 of study.

Prior Medication:

Allowed:

* Prior antiviral medication for HIV infection (if on such medication, must have received it for at least 2 weeks).
* Standard antimicrobial therapy for a documented positive gastrointestinal pathogen.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Gastrointestinal medications that cause diarrhea (e.g., magnesium-containing antacids, lactulose).
* Maintenance antifungal medication for life-threatening fungal infections (other than fluconazole <= 100 mg/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Surawicz CM, Study Chair
Locations (1):
- Madison Clinic, Seattle, Washington, United States

REFERENCES:
- [Background] McFarland LV, Surawicz CM, Greenberg RN, Fekety R, Elmer GW, Moyer KA, Melcher SA, Bowen KE, Cox JL, Noorani Z, et al. A randomized placebo-controlled trial of Saccharomyces boulardii in combination with standard antibiotics for Clostridium difficile disease. JAMA. 1994 Jun 22-29;271(24):1913-8. PMID 8201735